CLINICAL TRIAL: NCT05365126
Title: A Proof-of-concept Study of the Complete Vocal Technique (CVT), a Pedagogic Technique Used for Performers, in Improving the Voice and Vocal Function in Patients With Muscle Tension Dysphonia Using Telehealth
Brief Title: Complete Vocal Technique Voice Therapy for Muscle Tension Dysphonia (CVT4MTD)
Acronym: CVT4MTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19ET004
Record Dates: First submitted 2022-04-22; First posted 2022-05-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Muscle Tension Dysphonia
Keywords: Muscle Tension Dysphonia; Voice Therapy; Pilot study

STUDY DESIGN:
Intervention Model Description: Pilot/feasibility Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete Vocal Technique Voice Therapy (Experimental): Up to six 45 minute sessions delivered by a CVT Practitioner using a video link within an eight week therapy period
  Interventions: Behavioral: Complete Vocal Technique Voice Therapy

INTERVENTIONS:
Behavioral: Complete Vocal Technique Voice Therapy — A Complete Vocal Technique (CVT) Practitioner will assess the patient's voice and voice problems using the CVT framework and then apply CVT therapy, a form of voice therapy
  Other Names: CVT-VT

SUMMARY:
This proof-of-concept study is designed to evaluate whether a pedagogic technique used to help performers, known as the Complete Vocal Technique (CVT), can be used to help patients with a type of voice disorder known as Muscle Tension Dysphonia (MTD). MTD is responsible for up to 40% of patients presenting with voice and throat complaints. MTD is due to inefficient or ineffective voice production resulting from an imbalance in the control of the breathing mechanism, and uncontrolled constriction of the muscles in the larynx (voice box) or vocal tract (throat space above the vocal cords). Standard treatment is Voice Therapy delivered by a specialist Speech Therapist (SLT-V) often using a video link (telepractice aka telehealth). CVT is widely used in Europe by singers and vocal coaches. Practitioners (CVT- Ps) undergo a three-year accredited training programme, and the systematic and structured approach helps healthy singers and other performers optimise the function of the voice to produce any sound required. It also helps if the performer has vocal problems, which are also mainly due to uncontrolled throat constrictions.

The purpose of this pilot study is to see if the CVT voice therapy approach (CVT-VT) can help, and offers advantages, to standard SLT-V methods in the treatment of patients with MTD. Ten adult patients will be recruited from the Voice clinic at Nottingham University Hospital. Participants will have a multidimensional assessment using questionnaires, and voice recordings and then receive up to 6 video sessions of CVT-VT delivered using a video link by a CVT-P. The participants will then be reviewed back in clinic at 8 weeks and be reassessed, using further questionnaires and analysis of the voice pre- and post-therapy recordings, to evaluate the outcome of this treatment approach. Qualitative methodology will determine whether CVT-VT offers any therapeutic advantages to existing SLT-VT treatment methods.

DETAILED DESCRIPTION:
Voice problems (dysphonia) affect one in 13 adults annually, causes a major impact on quality of life and livelihood and is a substantial healthcare burden. It is more common in women and in those with vocally demanding professions and the elderly. Forty percent of patients referred for assessment of a voice problem have Muscle Tension Dysphonia (MTD) as a cause brought on by an imbalance of breathing mechanism and/or uncontrolled tightness of the muscles of the voice box or throat. The main symptoms are hoarseness, abnormal pitch or loudness, variability in quality or control of the voice, throat discomfort or difficulty in using the voice such as being able to use a louder voice when needed, or a voice that fatigues with use with a consequent impact on quality of life. Traditionally there are six described recognisable patterns of MTD based on the presenting symptoms, voice quality and on appearance of the larynx (voice box) on examination with a video camera. Three types (MTD patterns I-III) are more related to ineffective voice use, also known as 'voice abuse' or 'voice misuse', while the other three types (MTD patterns IV-VI) have a predominantly psychological basis.

In the United Kingdom (UK), patients with persistent or unexplained hoarseness who are over the age of 45 are referred under the two-week wait (2WW) cancer referral process. In other cases, referral to an Ear, Nose and Throat (ENT) benign voice service is usually considered if the dysphonia persists for more than six weeks, if it has not improved with simple measures such as voice rest, reducing irritation to the vocal cords and drinking plenty of fluids (known as vocal hygiene advice) or it is impacting significantly on the patient's work or social life. In practice patients with MTD may come through both the 2WW and benign voice pathways.

A diagnosis of MTD is made by an ENT surgeon and/or Speech & Language Therapist who has specialised in voice disorders (SLT-V) based on the history of the vocal complaint and by excluding an organic cause by examination of the patient's voice box (larynx) with a small flexible video camera passed through the nose. Treatment is with voice therapy given by a SLT-V. Voice therapy consists of two main types: Indirect Voice Therapy and Direct Voice Therapy and is guided by advice from professional organisations such as Royal College of Speech and Language Therapists Clinical Guidelines and the American Speech-Language-Hearing Association (ASHA) Clinical Practice Guideline: hoarseness (dysphonia). Indirect therapy consists of education, information, vocal hygiene, and stress management to encourage behavioural change. Direct therapy consists of establishing healthy voice production by rebalancing the three subsystems of voice production namely breathing (respiration), voice production (phonation) and more efficient use of resonance.

The aim of voice therapy is generally to (a) return the patient's voice to normal or as best as possible within the patient's anatomic and physiologic capabilities and (b) to satisfy the patient's occupational, social and emotional vocal needs and (c) promote habit changes that will ensure voice improvement will be maintained. Therapeutic goals should be specific and determined by the patient prior to therapy to empower the patient in shared decision making with the aim of improving motivation and compliance. In addition, the aim should be maximum improvement in the minimum time.

MTD is a mixed group of conditions with different patterns of presentation and numerous patient specific factors. In addition, Direct Voice Therapy is not just one treatment method and many SLT-Vs use a hierarchical approach, which focuses in the early stages on postural and relaxation techniques, followed by breathing exercises, voicing and resonance work with final consolidation and review. The techniques applied by a SLT-V are also dependent on abnormal findings on clinical examination the training and experience of the therapist and the response and engagement of the patient. Although having a large variety of techniques that can be used which can be tailored to the individual, Voice therapy has been portrayed as a "black box" and many recognised treatment regimens overlap in the treatment aims and therapeutic goals. This makes it difficult to determine why patients improve, which therapy tasks are most beneficial and for how long the tasks should be continued.

Another limitation of traditional Direct Voice Therapy can be that patients often have difficulty transferring the voice improvement on sustained vowels and during therapy sessions into conversational voice and day-to-day voice use. It is also recognised that patients do not always complete the therapy sessions in up to 18-65% of cases. Numerous reasons have been put forward for this, including clinician and clinic-related factors, gender, ethnicity, age, employment and perceived vocal severity, complex laryngeal diagnoses, additional medical problems, time commitment for treatment sessions or lack of rapid progress, adequate, if not complete, improvement in symptoms or failure to achieve goals. There is greater treatment satisfaction and likelihood of success if Direct Voice Therapy techniques are functionally orientated and have a more meaningful effect on quality of life with an emphasis on carryover activities into conversation so that it is more relevant to the patient's daily vocal demands. There is also increasing recognition that a patient may require more than one 'voice' to addresses the changing vocal needs (e.g., quiet talking, talking over noise, and yelling) in different environments.

Traditionally voice therapy has been given in a clinic environment face-to-face. However, with the onset of the Coronavirus (COVID-19) pandemic, Voice Therapy has almost entirely been given using telepractice via a video link. Prior to the COVID-19 pandemic, telepractice had been used by Speech and Language therapists mostly for geographical reasons and difficulties in patients' attending outpatient clinics. There are relatively few studies in its use for voice disorders and most studies on effectiveness have involved small cohorts of patients with a range of voice pathologies such as Parkinson's disease. There are few randomised controlled studies comparing face-to-face versus Telepractice and only one study of MTD patients using the same voice therapy technique (Flow phonation). This showed no significant difference in outcome between the two methods of delivery. Disadvantages of telepractice for voice therapy include generic problems with technology, patient environmental and cultural considerations, some instructional and practical issues with an inability to deliver more 'hands-on' techniques such as laryngeal manipulation. The Complete Vocal Technique (CVT) is pedagogic technique primarily used by singing teachers and vocal coaches to aid singers and actors produce the vocal sound and function that the performer requires. It has been used for over 35 years particularly in Europe and CVT practitioners (CVT-P) undergo an accredited 3-year training programme to achieve competency. It uses a hierarchical, systematic approach with terminology that is clearly defined and supported with scientific characterisation. It is based on four key building blocks enabling for example a singer to produce any vocal sound required in a healthy manner and regardless of genre of music. The first building block in CVT training is to ensure a healthy voice is produced by adopting the three overall principles: adequate support for the voice, use of a degree of twang ('necessary twang') and avoidance of jaw protrusion and tightening of the lips. Secondly one of four main vocal modes (Neutral, Curbing, Overdrive and Edge) is chosen which provides a set up for the larynx depending on the vocal requirement. These terms were introduced to avoid confusion with other more frequently used singing terms which lack precise definition. The choice of mode is determined by vocal demand (loudness, pitch range, vowel and genre 'norm' (vocal style) that is required: Neutral relates to normal conversational voice while the Curbing is a medium loud voice. Overdrive can be used for voice projection up to a shout loudness, while Edge can be used for a yelling and screaming quality. It would be expected that training in Neutral and Overdrive would allow good vocal function for most social situations for patients with MTD. The third element is to adjust the degree of sound colour (from dark to light) mostly achieved by lowering or raising the larynx and increasing or decreasing the pharyngeal space. The fourth element is to add specific vocal effects such as vibrato, ornamentation, distortion etc., which can be added once the first three have been achieved. In this way the precise sound required by the singer can be fashioned in any style or genre of music. The principles have been applied to training the speaking voice and provide a recipe for producing any desired voice quality for any environmental situation. A similar approach, that has not been widely adopted, has also been described whereby the aim is not to support the production of 'one voice', as is frequently the case with traditional SLT-VT, but to provide the patient with a range of 'new' voices to meet the patient's vocal needs.

Training programmes have been developed, using this methodology, to enable singers and singing teachers to improve, achieve vocal goals and overcome technical issues many of which are due to unintentional hyper-constrictive muscle activity within the larynx and vocal tract. CVT has also been applied to problems with the professional speaking voice and can help with reducing constriction and improved voice production and projection. Specific elements of CVT have also been packaged together in what is termed CVT Voice Therapy (CVT-VT). CVT-VT is used for singers and other performers presenting with acute vocal problems leading to hoarseness or loss of voice when time is of the essence in getting a vocalist back to professional voice use. Although widely used by CVT-Ps and published in several books it has not been formally evaluated.

The application of telepractice during the COVID-19 pandemic has also become a necessity in teaching singing and has been adopted by the Complete Vocal Institute (CVI) in Denmark where almost all tuition is now delivered on-line. Informal feedback from singers has been positive with many advantages (comfort of own home, reduction in cost, and no travel time) outweighing the disadvantages (some technical issues with audio/connection). It is likely a complete return to previous methods of delivery of SLT and CVT practice will not happen after the COVID-19 pandemic with the adoption of the new methods of service delivery for both.

In conclusion, the rationale for this Proof-of Concept study is to see whether an established pedagogic technique, CVT, which is used to train singers and performers with healthy voices and restore the voice when not functioning, can be used to treat patients with MTD and whether it offers advantages to traditional SLT-VT techniques. Many of the voice problems in performers and patients are due to faulty technique of voice production and are therefore similar to patients with MTD. In addition, the focus of CVT is not only to improve the voice and vocal function by reducing unhealthy throat constrictions but also allowing patients to develop the voice needed for the vocal requirement. Further, the terms and pedagogic process used in CVT are well defined and the theoretical framework on which it is built has been extensively investigated. The main questions are does it offer benefit, and how does it differ, from traditional SLT-VT methods and could it be a useful additional tool for SLT-VTs in the management of MTD?

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary Muscle Tension Dysphonia (MTD) based on history and laryngoscopic assessment (Type (I-III) MTD pattern) through joint assessment by a SLT-V and laryngologist
* Current voice problems, persistent for greater than 2 months
* Severity of disorder a) Voice Handicap Index (VHI) ≥ 30 and b) patient wants therapy
* Patient willingness to undergo treatment
* Consent to participate in study protocol

Exclusion Criteria:

* Organic vocal pathology 1) Structural/neoplastic disorders (e.g. carcinoma, cyst, polyp, papilloma, Reinke's oedema); 2) neurological disorders (e.g. vocal cord palsy, paresis, spasmodic dysphonia); 3) inflammation (e.g. infection, reflux (RFS >7) or significant relevant systemic disease (e.g. severe Chronic Obstructive Pulmonary Disease) or need for surgery
* Significant psychological issues identified during initial assessment (with option to withdraw if discovered during the treatment periods and agreed by both patient and Therapist)
* MTD pattern (IV-VI) compatible with significant primary psychological aetiology on laryngoscopy
* Transgender voice issues
* Previously incompletely treated dysphonia, neurological disease, or upper aerodigestive tract malignancy Had previous Voice Therapy (VT) or CVT training or pharmacological treatment for their voice problem - (other than proton pump inhibitors or an alginate recommended for disorders of laryngopharyngeal reflux-related symptoms)
* A hearing impairment that would prohibit or impact on telepractice treatment
* Significant concomitant health problems affecting voice
* Not have or be able to use a computer with video link at home or in hospital even with support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index (VHI) | Eight weeks
  Questionnaire to evaluate patient's self-reported perception of the impact of his or her voice disorder

SECONDARY OUTCOMES:
Patient Experience Feedback Form: Achievement of specific goals | Eight weeks
  Questionnaire to evaluate the patient defined goals of treatment defined pre-treatment and agreed with CVT practitioner
Patient Experience Feedback Form: Experience of therapy | Eight weeks
  Questionnaire to evaluate the patient's perception of satisfaction with therapy
CVT Practitioner Experience Feedback Form: Achievement of specific goals | Eight weeks
  Questionnaire to evaluate the CVT Practitioner's perception of achievement of defined goals of treatment defined pre-treatment and agreed with patient
CVT Practitioner Experience Feedback Form: Experience of therapy | Eight weeks
  Questionnaire to evaluate the CVT Practitioner's perception of Complete Vocal Technique (CVT) therapy for the patient
Feedback form: use of the video link | Eight weeks
  Questionnaire to evaluate the use of the video link by both the patient and CVT Practitioner
Acoustic and Electroglottographic (EGG) voice analysis pre and pots-therapy | Eight weeks
  A range of simultaneously acquired acoustic and EGG measures made on voice recordings of continuous speech, phrases based on phonetically selected texts and sustained vowels
Psychoacoustic evaluation of the recorded voice samples | Eight weeks
  The Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) and a CVT derived assessment tool will be used to demonstrate whether there is a perceptual change in the voice and which specific parameters have changed
Vocal tract discomfort scale questionnaire | Eight weeks
  A self-reported rating scale questionnaire which allows the patient to rate the frequency and severity of eight items pre- and post therapy
The Maximum Phonation Time (MPT) | Eight weeks
  An aerodynamic measure of the ability to sustained a vowel. This will be tested pre- and post-therapy

OTHER OUTCOMES:
Qualitative comparison of the specific techniques used by the CVT Practitioner compared to standard Speech Therapy techniques | Eight weeks
  Qualitative assessment based on a log of techniques used during the therapy session and qualitative assessment of anonymised, redacted transcripts of therapy sessions in those who have given additional consent

CONTACTS AND LOCATIONS:
Overall Officials: Julian A McGlashan, FRCS(Otol.), Principal Investigator — Nottingham University Hospitals; Cathrine Sadolin, Study Director — Complete Vocal Institute
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGlashan J, Aaen M, White A, Saccente-Kennedy B, Tempesta M, Sadolin C. Feasibility and Acceptability of Complete Vocal Technique-Voice Therapy as a Treatment for Primary Muscle Tension Dysphonia: A Feasibility Trial. J Voice. 2025 Sep 4:S0892-1997(25)00308-X. doi: 10.1016/j.jvoice.2025.07.044. Online ahead of print. PMID 40913007
- [Derived] McGlashan J, Aaen M, White A, Sadolin C. A mixed-method feasibility study of the use of the Complete Vocal Technique (CVT), a pedagogic method to improve the voice and vocal function in singers and actors, in the treatment of patients with muscle tension dysphonia: a study protocol. Pilot Feasibility Stud. 2023 May 24;9(1):88. doi: 10.1186/s40814-023-01317-y. PMID 37226281
- See also: Protocol publication — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-023-01317-y

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT05365126/Prot_SAP_ICF_000.pdf